CLINICAL TRIAL: NCT04813666
Title: Role of Detection of Lipoarabinomannan (LAM) in Urine for Diagnosis of Pulmonary Tuberculosis in HIV Patients; Egyptian Experience
Brief Title: Lipoarabinomannan (LAM) in Urine for Diagnosis of Pulmonary Tuberculosis in HIV Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Assem Hewidy, assistant professor of chest medicine, Mansoura University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: MansouraU LAM
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: TB - Tuberculosis HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TB group (Active Comparator)
  Interventions: Diagnostic Test: Urinary LAM ELISA:
- Non TB group (Placebo Comparator)
  Interventions: Diagnostic Test: Urinary LAM ELISA:

INTERVENTIONS:
Diagnostic Test: Urinary LAM ELISA:

SUMMARY:
A diagnostic validity study in which urinary LAM was done in seropositive HIV patients with symptoms suggestive of TB who were included and investigated with battery of tests to reach the final diagnosis.

DETAILED DESCRIPTION:
A diagnostic validity study in which urinary LAM was done in seropositive HIV patients with symptoms suggestive of TB who were included and investigated with battery of tests to reach the final diagnosis.

The study was conducted at Mansoura Fever Hospital in collaboration with the Chest Department and Clinical Pathology Department, Mansoura University, Egypt, from January 2015 to October 2016.

Ethical approval had been obtained from Medical Research Ethics Committee of Faculty of Medicine, Mansoura University (code no: MD/138). Approval from Egyptian Ministry of Health was taken (No: 1-2016/18). Patients signed their written consents after detailed explanation of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* The study included seropositive HIV patients with a new diagnosis of either pulmonary or extra-pulmonary TB, and also included patients who were presented by symptoms suggestive for tuberculosis, changes in chest X ray that not improved by full course of antibiotics or positive tuberculin test ≥ 5 mm.

Exclusion Criteria:

* Patients on anti-TB drugs or negative screening for sero-positive HIV patients were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
positive for TB | day 1
  Concentration of urinary LAM was done in seropositive HIV patients

IPD SHARING:
Plan to Share IPD: No
NO plan